CLINICAL TRIAL: NCT00576134
Title: Artificial Larynx : Intralaryngeal Prosthesis With Valve in Major Swallowing Troubles
Brief Title: The Objective is to Respond to Patients' Needs in the Field of Larynx Replacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3866
Record Dates: First submitted 2007-12-12; First posted 2007-12-18 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Swallowing Disorders; Dysphagia; Laryngeal Neoplasms
Keywords: Larynx, tracheotomy, titanium beads
MeSH Terms: conditions — Deglutition Disorders; Laryngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantation of intralaryngeal prosthesis with a new double valve system, allowing tracheotomy closing — An artificial Larynx composed of a tracheobronxane ® Dumon ST prosthesis and a valves system will be implant under general anesthesia by endoscopy. The 3 first patients will be patients with tracheotomy, in order to allow breathing through this tracheotomy in case of valves dysfunction.

SUMMARY:
Supplement pharyngolaryngeal deficient functions by insertion of a prosthesis with valves in order to allow tracheotomy closing (when applicable) and / or to allow restoration of god swallowing capacity. The secondary objective is to study the concept of a special valves system for the development of an artificial larynx

ELIGIBILITY:
Inclusion criteria:

* Age more than 18
* Swallowing troubles

Exclusion criteria:

* Pregnant women
* Contraindications to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Respiratory evaluation | Day : 1, 2, 3, 4, 5, 15 - month :1, 3, 6, 12, 18, 24, 30, 36

SECONDARY OUTCOMES:
Nasofibroscopy | Day : 15 - month : 1, 3, 6, 12, 18, 24, 30, 36

CONTACTS AND LOCATIONS:
Overall Officials: Christian DEBRY, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale, Hôpital de Hautepierre, 1 avenue Molière, Strasbourg, France

REFERENCES:
- [Result] Chambres O, Schultz P, Debry C. The Larynxane ST intralaryngeal endoprosthesis for laryngotracheal pathologies. J Laryngol Otol. 2006 Nov;120(11):942-8. doi: 10.1017/S0022215106000466. Epub 2006 May 4. PMID 16672085
- [Result] Debry C, Charles X, Frenot M, Gentine A. Intra-laryngeal endoprosthesis: an alternative therapeutic approach to surgical procedures of laryngeal exclusion. J Laryngol Otol. 2000 Oct;114(10):760-4. doi: 10.1258/0022215001904095. PMID 11127145